CLINICAL TRIAL: NCT05453279
Title: A Single and Multiple Dose Escalation First-In-Human Study Evaluating the Safety, Tolerability, and Pharmacokinetics of Delcetravir Administered Via Inhalation in Healthy Subjects
Brief Title: A Dose Escalation Phase 1 Study Evaluating the Safety and Pharmacokinetics of an Inhaled COVID-19 Inhibitor Delcetravir in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Esfam Biotech Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COV0001
Record Dates: First submitted 2022-06-01; First posted 2022-07-12 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This study will be a single center, Phase I, randomized, double-blind, placebo controlled, single and multiple ascending dose (SAD/MAD) study evaluating safety, tolerability, and PK after administration via oral inhalation in healthy subjects.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind allocation to inhalation formulation (active or placebo)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (experimental) (Active Comparator): Delcetravir inhalation via dry powder inhaler device administered up to 4 single ascending doses. According to tolerability of single ascending doses, delcetravir is then given as inhalation via dry powder device in multiple ascending doses, once daily for 7 days.
  Interventions: Combination Product: Delcetravir dry powder inhaler
- Placebo comparator (Placebo Comparator): Placebo inhaler, identical in appearance to the active comparator, administered doses up to 4 single ascending doses. According to tolerability of single ascending doses, placebo doses are then given as inhalation via dry powder device in multiple ascending doses, once daily for 7 days.
  Interventions: Combination Product: Delcetravir dry powder inhaler

INTERVENTIONS:
Combination Product: Delcetravir dry powder inhaler — Placebo dry powder inhaler

SUMMARY:
This study will be a single center, Phase I, randomized, double-blind, placebo controlled, single and multiple ascending dose (SAD/MAD) study evaluating the safety, tolerability, and PK of Delcetravir after administration via oral inhalation in healthy subjects.

DETAILED DESCRIPTION:
Primary objectives:

* To evaluate the safety and tolerability of single and multiple doses of Delcetravir in healthy subjects (18-50 years of age).
* To evaluate the safety and tolerability of single and multiple doses of Delcetravir in healthy subjects (50-80 years of age).
* To evaluate the pharmacokinetics (PK) of Delcetravir after single and multiple doses of ESFAM289 in healthy subjects (18-50 years of age).
* To evaluate the PK of Delcetravir after single and multiple doses of Delcetravir in healthy subjects (50-80 years of age)

Secondary objectives:

* To compare the PK of Delcetravir after single and multiple doses of Delcetravir in age stratified subjects (18-50 vs. 50-80 years of age).
* To compare the safety and tolerability after single and multiple doses of Delcetravir in age stratified subjects (18-50 vs. 50-80 years of age).

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be included in the study:

1. Male or female, non-smokers or casual smokers (defined as smoking the equivalent of less than an average of 5 cigarettes per week, and willing to abstain from smoking during involvement in the study), ≥18 and <50 (For Parts A and B) or ≥50 and ≤80 (for Parts C and D) years of age, with BMI >18.0 and <32.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
2. Healthy as defined by:

   1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
   2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Females of childbearing potential who are sexually active with a male partner must be willing to use one of the following acceptable contraceptive methods throughout the study and for 30 days after the last study drug administration:

   1. Simultaneous use of intra-uterine device placed at least 4 weeks prior to study drug administration, and condom for the male partner;
   2. Simultaneous use of hormonal contraceptives started at least 4 weeks prior to study drug administration and condom for the male partner.
   3. Sterile male partner (vasectomized since at least 6 months).
4. Females of non-childbearing potential must be:

   1. Post-menopausal (defined as absence of menses for at least 12 months prior to the first study drug administration) with confirmation of the post menopausal status by documented FSH level greater than 40 mIU/mL; or
   2. Surgically sterile (complete hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or tubal ligation at least 6 months prior to the first study drug administration).
5. Male subjects who are not vasectomized for at least 6 months, and who are sexually active with a female partner of childbearing potential (childbearing potential females are defined as women that are neither post-menopausal nor surgically sterile) must be willing to use one of the following acceptable contraceptive methods from the first study drug administration until at least 90 days after the last study drug administration:

   a) Simultaneous use of a male condom and, for the female partner, hormonal contraceptives used since at least 4 weeks, or intra-uterine contraceptive device placed since at least 4 weeks;
6. Male subjects who are sexually active with a same-sex partner must be willing to use a condom until study exit.
7. Male and female subjects who practice abstinence from sexual intercourse as a usual and preferred lifestyle.
8. Male subjects must be willing not to donate sperm until 90 days following the last study drug administration.
9. Subjects with normal lung function defined as ≥80% predicted forced expiratory volume in one second (FEV1) at screening.
10. Capable of consent.

Exclusion criteria:

1) Any clinically significant abnormality at physical examination, clinically significant abnormal laboratory test results or positive test for HIV, hepatitis B, or hepatitis C found during medical screening.

2) Any clinically significant illness, infection, medical/surgical procedure, or trauma within 4 weeks of check-in, or planned inpatient surgery or hospitalization during the study period.

3) Any history of malignancy or neoplastic disease

1. Positive urine drug screen, urine cotinine test, or alcohol breath test at screening.
2. History of significant allergic reactions (e.g., drug reaction, anaphylactic reaction, hypersensitivity, angioedema) to any drug.
3. Positive pregnancy test at screening.
4. Clinically significant ECG abnormalities (QTc greater than 450 ms) or vital sign abnormalities (systolic blood pressure less than 90 or greater than140 mmHg, diastolic blood pressure less than 40 or greater than 90 mmHg, or heart rate less than 40 or greater than100 bpm, oxygen saturation less than 95% O2) at screening.
5. History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to the screening visit. Regular use of alcohol is defined as greater than 14 units of alcohol per week, where 1 unit is defined as 375 mL of beer at 3.5% a/v, 100 mL of wine at 13.5% a/v, or 30 mL of spirit at 40% a/v.
6. History of drug abuse within 1 year prior to screening, recreational use of soft drugs (such as tetrahydrocannabinol [THC]) within 1 month prior to the screening visit, or hard drugs (amphetamines, methamphetamines, methadone, barbiturates, benzodiazepines, cocaine, opiates, methyledioxymethamphetamine [MDMA], and phencyclidine [PCP]) within 3 months prior to screening.
7. Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing, or concomitant participation in an investigational study involving no drug or device administration.
8. Use of medications for the timeframes specified below, with the exception of medications exempted by the Investigator on a case-by-case basis because they are judged unlikely to affect the PK profile of the study drug or subject safety (e.g., topical drug products without significant systemic absorption):

   1. Prescription medications (except for hormonal contraceptives) within 14 days prior to the first dosing;
   2. Over-the-counter products and natural health products (including herbal remedies, such as St. John's wort, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports) within 7 days prior to the first dosing, with the exception of the occasional use of acetaminophen/paracetamol (up to 2 g/day), ibuprofen (up to 800 mg/day), and topical formulations without significant systemic absorption;
   3. Depot injection or implant (except for hormonal contraceptives) of any drug within 3 months prior to the first dosing.
9. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to the first dosing.
10. Breast-feeding subject.
11. History of latent or active tuberculosis, or exposure to endemic areas within 8 weeks prior to QuantiFERON®-TB testing performed at screening.
12. Positive QuantiFERON®-TB test indicating possible tuberculosis infection.
13. Immunization with a live attenuated vaccine within 1 month prior to dosing or planned vaccination during the course of the study.
14. Presence of fever (body temperature greater than 37.6 °C) e.g. a fever associated with a symptomatic viral or bacterial infection, within 2 weeks prior to the first dosing.
15. Any reason that, in the opinion of the Investigator, would prevent the subject from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with chest pain after single and multiple ascending doses of active and placebo comparator | 22 days
  Symptoms of chest pain
Number of subjects with shortness of breath after single and multiple ascending doses of active and placebo comparator | 22 days
  Symptoms of shortness of breath
Number of subjects with cough after single and multiple ascending doses of active and placebo comparator | 22 days
  Symptoms of cough
Number of subjects with sputum production after single and multiple ascending doses of active and placebo comparator | 22 days
  Symptoms of sputum production
Hemoglobin assessment after active comparator and placebo. | 22 days
  Hemoglobin in g/L
White cell count assessment after active comparator and placebo. | 22 days
  White cell count differential in 109/L
Platelet count assessment after active comparator and placebo. | 22 days
  Platelet count in 109/L
Laboratory meaurement of sodium concentration after active comparator and placebo. | 22 days
  Serum sodium in mmol/L
Laboratory measurement of potassium concentration after active comparator and placebo. | 22 days
  Serum potassium in mmol/L
Laboratory measurement of bicarbonate concentration after active comparator and placebo. | 22 days
  Serum bicarbonate in mmol/L
Laboratory measurement of urea concentration after active comparator and placebo. | 22 days
  Serum urea in mmol/L
Laboratory measurement of creatinine concentration after active comparator and placebo. | 22 days
  Serum creatinine in umol/L
Laboratory measurement of ALT concentration after active comparator and placebo. | 22 days
  Serum ALT in U/L
Laboratory measurement of AST concentration after active comparator and placebo. | 22 days
  Serum AST in U/L
Laboratory measurement of alkaline phosphatase concentration after active comparator and placebo. | 22 days
  Serum alkaline phosphatase in U/L
Heart rate after active comparator and placebo. | 22 days
  Heart rate in beats per minute
Blood pressure after active comparator and placebo. | 22 days
  Systolic and diastolic blood pressure in mmHg
Respiratory rate after active comparator and placebo. | 22 days
  Respiratory rate in breaths per minute
Pulse oximetry measurement after active comparator and placebo. | 22 days
  Pulse oximetry in blood oxygen saturation
ECG after active comparator and placebo. | 22 days
  PR interval, QRS complex, QTc interval

CONTACTS AND LOCATIONS:
Overall Officials: Albert G Frauman, MD, Study Director — Esfam Biotech Pty Ltd

IPD SHARING:
Plan to Share IPD: No